CLINICAL TRIAL: NCT00457912
Title: Genetic Characterization of Individuals With Limb Girdle Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Jerry R. Mendell, DIRECTOR CENTER FOR GENE THERAPY, Nationwide Children's Hospital
Other Study IDs: IRB05-00101; NIH Grant U54AR050733
Record Dates: First submitted 2007-04-06; First posted 2007-04-09 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Limb-Girdle Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, muscle tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to identify and maintain a registry of well-characterized limb-girdle muscular dystrophy (LGMD) patients. Patients seen as part of this study may be candidates for future treatment trials based on their defined genetic classification of LGMD. In the course of this study, the investigators will perform a muscle biopsy and DNA testing in an unlimited number of patients with clinically diagnosed LGMD. The genetic testing will be extended to the family of the study subject in order to better understand true genetic defect.

ELIGIBILITY:
Inclusion Criteria:

* any subject with clinical diagnosis of LGMD
* must visit Columbus Children's Hospital for 2-day study visit
* muscle biopsy tissue must be available; either from previous biopsy, affected relative, or willing to have biopsy at Columbus Children's

Exclusion Criteria:

* diagnosis of a neuromuscular disorder other than LGMD
* unable to provide muscle tissue from previous or current biopsy
* incapable of giving consent and not having a legal guardian willing or able to do so

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any subject with clinical diagnosis of LGMD
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2005-06; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R. Mendell, M.D., Principal Investigator — The Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States